CLINICAL TRIAL: NCT02200315
Title: Phase II Study of the Efficacy of no Antimicrobial Prophylaxis Use for Laparoscopic Distal Gastrectomy for Gastric Carcinoma
Brief Title: No Antimicrobial Prophylaxis for Laparoscopic Distal Gastrectomy
Acronym: KSWEET-01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Korean South West East Gastric Surgery Group (Other)
Responsible Party: Principal Investigator, Oh Jeong, Associate Professor, Korean South West East Gastric Surgery Group
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSWEET-01
Record Dates: First submitted 2014-07-21; First posted 2014-07-25 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Stomach Neoplasms
Keywords: Stomach neoplasms; Surgical site infection; Laparoscopic gastrectomy; Antimicrobial prophylaxis
MeSH Terms: conditions — Stomach Neoplasms; Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- No Antimicrobial prophylaxis (Experimental): No use of antimicrobial prophylaxis during surgery
  Interventions: Other: No Antimicrobial prophylaxis

INTERVENTIONS:
Other: No Antimicrobial prophylaxis — Antimicrobial prophylaxis are not administered during an operation

SUMMARY:
The aim of this study is to evaluate the feasibility and safety of no use of antimicrobial prophylaxis during laparoscopic distal gastrectomy for gastric carcinoma.

DETAILED DESCRIPTION:
This is a phase II clinical trial investigating the postoperative surgical site infection (SSI) rates after no antimicrobial prophylaxis use during laparoscopic distal gastrectomy. Target ranges of SSI rates after laparoscopic distal gastrectomy were determined based on the previous reports and our data. If SSI rates are within the target range, the investigators will proceed to a randomized controlled trial investigating the efficacy of no antimicrobial use for laparoscopic gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven gastric adenocarcinoma clinical stage T1-2N0M0 patients who underwent laparoscopic distal gastrectomy
* Age between 18 and 65 years
* American Society of Anaesthesiologists (ASA) status >2
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Normal blood, liver, pulmonary, cardiac, and renal function
* Informed consent

Exclusion Criteria:

* Administration of antibiotics within 1 month before surgery
* Active infection at the time of surgery
* Combined resection during operation (i.e., spleen, liver, colon, etc.)
* History of upper abdominal surgery
* Previous chemotherapy or radiotherapy within 6 months before surgery
* Uncontrolled underlying comorbidities
* Malnutrition with BMI less than 18.5 kg/m2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2014-05; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Postoperative surgical site infection | Within postoperative 1 month
  Incidence of surgical site infection, including superficial incisional, deep incisional, and organ/space infection, until postoperative 1 month

SECONDARY OUTCOMES:
Postoperative morbidity and mortality | Within postoperative 1 month or during hospitalization
  Occurence of postoperative complications or deaths until postoperative 1 months or during hospitalization. Postoperative complications will be assessed with respect to types and severity.
Hospital stay | Up to 1month after operation
  The duration of hospital stay from the operation to hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Oh Jeong, MD, PhD, Study Director — Chonnam National University Hospital; Young Kyu Park, MD, PhD, Study Chair — Chonnam National University Hospital
Locations (3):
- South Korea (3):
  - Chonnam National University Hwasun Hospital, Hwasun-eup, Jeollanam-do
  - Dong-A University Hospital, Busan, Kyungsang-do
  - Kyemyung University Dongsan Medical Center, Daegu, Kyungsang-do

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burke JP. Infection control - a problem for patient safety. N Engl J Med. 2003 Feb 13;348(7):651-6. doi: 10.1056/NEJMhpr020557. No abstract available. PMID 12584377
- [Background] Choudhary A, Bechtold ML, Puli SR, Othman MO, Roy PK. Role of prophylactic antibiotics in laparoscopic cholecystectomy: a meta-analysis. J Gastrointest Surg. 2008 Nov;12(11):1847-53; discussion 1853. doi: 10.1007/s11605-008-0681-x. Epub 2008 Sep 9. PMID 18780131
- [Background] McDonald M, Grabsch E, Marshall C, Forbes A. Single- versus multiple-dose antimicrobial prophylaxis for major surgery: a systematic review. Aust N Z J Surg. 1998 Jun;68(6):388-96. doi: 10.1111/j.1445-2197.1998.tb04785.x. PMID 9623456
- [Background] Bratzler DW, Dellinger EP, Olsen KM, Perl TM, Auwaerter PG, Bolon MK, Fish DN, Napolitano LM, Sawyer RG, Slain D, Steinberg JP, Weinstein RA; American Society of Health-System Pharmacists; Infectious Disease Society of America; Surgical Infection Society; Society for Healthcare Epidemiology of America. Clinical practice guidelines for antimicrobial prophylaxis in surgery. Am J Health Syst Pharm. 2013 Feb 1;70(3):195-283. doi: 10.2146/ajhp120568. No abstract available. PMID 23327981
- [Background] Imai E, Ueda M, Kanao K, Miyaki K, Kubota T, Kitajima M. Surgical site infection surveillance after open gastrectomy and risk factors for surgical site infection. J Infect Chemother. 2005 Jun;11(3):141-5. doi: 10.1007/s10156-005-0379-x. PMID 15990978
- [Background] Imamura H, Furukawa H, Iijima S, Sugihara S, Tsujinaka T, Tsukuma H, Shimokawa T. Multicenter phase II study of antimicrobial prophylaxis in low-risk patients undergoing distal gastrectomy for gastric cancer. Gastric Cancer. 2006;9(1):32-5. doi: 10.1007/s10120-005-0354-3. PMID 16557434
- [Background] Migita K, Takayama T, Matsumoto S, Wakatsuki K, Enomoto K, Tanaka T, Ito M, Nakajima Y. Risk factors for surgical site infections after elective gastrectomy. J Gastrointest Surg. 2012 Jun;16(6):1107-15. doi: 10.1007/s11605-012-1838-1. Epub 2012 Feb 15. PMID 22350727
- [Background] Memon MA, Khan S, Yunus RM, Barr R, Memon B. Meta-analysis of laparoscopic and open distal gastrectomy for gastric carcinoma. Surg Endosc. 2008 Aug;22(8):1781-9. doi: 10.1007/s00464-008-9925-9. Epub 2008 Apr 25. PMID 18437472
- [Background] Kim HH, Hyung WJ, Cho GS, Kim MC, Han SU, Kim W, Ryu SW, Lee HJ, Song KY. Morbidity and mortality of laparoscopic gastrectomy versus open gastrectomy for gastric cancer: an interim report--a phase III multicenter, prospective, randomized Trial (KLASS Trial). Ann Surg. 2010 Mar;251(3):417-20. doi: 10.1097/SLA.0b013e3181cc8f6b. PMID 20160637
- [Background] Ammori BJ. A prospective randomized study of prophylactic antibiotics in elective laparoscopic cholecystectomy. Surg Endosc. 2004 Mar;18(3):565; author reply 566. doi: 10.1007/s00464-003-9141-6. Epub 2004 Feb 2. No abstract available. PMID 14973693
- [Background] Catarci M, Mancini S, Gentileschi P, Camplone C, Sileri P, Grassi GB. Antibiotic prophylaxis in elective laparoscopic cholecystectomy. Lack of need or lack of evidence? Surg Endosc. 2004 Apr;18(4):638-41. doi: 10.1007/s00464-003-9090-0. Epub 2004 Feb 2. PMID 14752639
- [Background] Culver DH, Horan TC, Gaynes RP, Martone WJ, Jarvis WR, Emori TG, Banerjee SN, Edwards JR, Tolson JS, Henderson TS, et al. Surgical wound infection rates by wound class, operative procedure, and patient risk index. National Nosocomial Infections Surveillance System. Am J Med. 1991 Sep 16;91(3B):152S-157S. doi: 10.1016/0002-9343(91)90361-z. PMID 1656747
- [Derived] Jeong O, Jung MR, Ryu SY, Park YK, Kim MC, Kim KH, Ryu SW, Kwon IG, Son YG. Multicenter Phase 2 Study about the Safety of No Antimicrobial Prophylaxis Use in Low-Risk Patients Undergoing Laparoscopic Distal Gastrectomy for Gastric Carcinoma (KSWEET-01 Study). Gastroenterol Res Pract. 2017;2017:8928353. doi: 10.1155/2017/8928353. Epub 2017 Jun 5. PMID 28656047